CLINICAL TRIAL: NCT03485287
Title: An Open-Label, Multi-Site Phase 2 Study of the Safety and Effect of Manualized MDMA-Assisted Psychotherapy for the Treatment of Severe Posttraumatic Stress Disorder (Canada)
Brief Title: Study of Safety and Effects of MDMA-assisted Psychotherapy for Treatment of PTSD (Canada)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lykos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP-17
Record Dates: First submitted 2018-03-23; First posted 2018-04-02 (Actual); Results first posted 2021-07-01 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; MDMA; Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Intervention Model Description: Three sessions of MDMA-assisted therapy with flexible dose of MDMA (100 to 125 mg with optional supplemental half-dose)
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- MDMA-assisted therapy (Experimental): Three sessions of MDMA-assisted therapy with flexible dose of midomafetamine HCl from 100 to 125 mg and optional supplemental dose half that of initial dose 1.5 to 2 hours later
  Interventions: Drug: Midomafetamine HCl; Behavioral: Manualized therapy

INTERVENTIONS:
Drug: Midomafetamine HCl — Three sessions of MDMA-assisted therapy with flexible dose of midomafetamine HCl from 100 to 125 mg and optional supplemental dose half that of initial dose 1.5 to 2 hours later
  Other Names: 3,4-methylenedioxymethamphetamine; MDMA; MDMA HCl; midomafetamine
Behavioral: Manualized therapy — Non-directive therapy

SUMMARY:
The goal of this clinical trial is to learn if MDMA-assisted therapy is safe and effective at reducing PTSD symptoms in people with at least severe PTSD.

The main question it aims to answer is:

Do three open-label sessions of MDMA-assisted therapy reduce PTSD symptoms?

Participants will receive three non-drug preparatory sessions followed by three sessions of MDMA-assisted therapy. Each MDMA-assisted therapy session is followed by three non-drug integrative therapy sessions.

DETAILED DESCRIPTION:
This multi-site, open-label, Phase 2, lead-in study assesses the safety and effect of MDMA-assisted therapy in participants diagnosed with at least severe posttraumatic stress disorder (PTSD). Therapy teams that have been identified and trained to work on the sponsor's planned Phase 3 studies will treat at least one open-label participant in this study.

This study will compare the effects of three open-label manualized Experimental Sessions of psychotherapy assisted by flexible doses of MDMA. Initial doses per Experimental Session include 100 mg or 125 mg of MDMA compounded with lactose, followed 1.5 to 2 hours later by a supplemental half-dose (50 mg or 62.5 mg). Total amounts of MDMA to be administered per Experimental Session range from 100 mg to 187.5 mg. This ~12-week Treatment Period is preceded by three Preparatory Sessions. During the Treatment Period, each Experimental Session is followed by three Integrative Sessions of non-drug psychotherapy.

The primary outcome measure is the change in the Clinician Administered PTSD Scale for DSM 5 (CAPS-5) total severity scores from Baseline to Visit 19. The secondary outcome measure is the change in the customized version of the Sheehan Disability Scale (SDS) for PTSD for the MAPS studies total scores from Baseline to Visit 19.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years old
* Are fluent in speaking and reading the predominantly used or recognized language of the study site
* Agree to have study visits recorded, including Experimental Sessions, Independent Rater assessments, and non-drug psychotherapy sessions
* Must provide a contact (relative, spouse, close friend or other caregiver) who is willing and able to be reached by the investigators in the event of a participant becoming suicidal or unreachable.
* Must agree to inform the investigators within 48 hours of any medical conditions and procedures.
* If of childbearing potential, must have a negative pregnancy test at study entry and prior to each Experimental Session, and must agree to use adequate birth control through 10 days after the last Experimental Session.
* Must not participate in any other interventional clinical trials during the duration of the study,
* Must be willing to remain overnight at the study site after each Experimental Session and be driven home after, and commit to medication dosing, therapy, and study procedures

Exclusion Criteria:

* Are not able to give adequate informed consent
* Have uncontrolled hypertension
* Have a marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 milliseconds [ms] corrected by Bazett's formula)
* Have a history of additional risk factors for Torsade de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
* Have evidence or history of significant medical disorders
* Have symptomatic liver disease
* Have history of hyponatremia or hyperthermia
* Weigh less than 48 kilograms (kg)
* Are pregnant or nursing, or are of childbearing potential and are not practicing an effective means of birth control.
* Meet DSM-5 criteria for active substance use disorder for any substance other than caffeine or nicotine
* Have used Ecstasy (material represented as containing MDMA) more than 10 times within the last 10 years or at least once within 6 months of the first Experimental Session; or have previously participated in a MAPS or Lykos-sponsored MDMA clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2019-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mithoefer, Study Director — MAPS Public Benefit Corp.
Locations (2):
- Canada (2):
  - British Columbia Centre on Substance Abuse, Vancouver, British Columbia
  - Dr. Simon Amar, LLC, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
We will share outcome data appearing in any published reports upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data and study-related documents will be available when all participants have completed the study
Access Criteria: Interested persons should correspond with the central contact for study.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants will be recruited through print and internet advertisements, referrals from other psychiatrists, psychotherapists, or physicians, and by word of mouth.
Groups:
- MDMA-assisted Therapy (100 to 125 mg): Three sessions of open-label MDMA-assisted therapy with flexible dose of midomafetamine HCl from 100 to 125 mg and optional supplemental dose half that of initial dose 1.5 to 2 hours later
Period: Overall Study
Arm/Group | MDMA-assisted Therapy (100 to 125 mg)
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety Set
Arm/Group | MDMA-assisted Therapy (100 to 125 mg)
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.25 (5.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Disabled from Work [Count of Participants; unit: Participants]
  Yes | 1
  No | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Primary Endpoint in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Severity Score
Description: The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) is a clinician administered and scored assessment of PTSD symptoms via structured interview based upon PTSD diagnosis in DSM-5. It contains symptom subscales, a CAPS-5 total severity score, and a diagnostic score. The total severity score is a sum of symptom frequency and intensity scores for the subscales B (re-experiencing), C (avoidance) and D (hypervigilance) and ranges from 0 to 136, with higher scores indicating greater severity of PTSD symptoms.
Time Frame: Baseline (Visit 3) to Primary Endpoint (Visit 19,18 weeks post enrollment)
Population: Safety Set
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- MDMA-assisted Therapy (100 to 125 mg of MDMA): Three sessions of open-label MDMA-assisted therapy with flexible dose of MDMA from 100 to 125 mg and optional supplemental dose half that of initial dose 1.5 to 2 hours later.
Arm/Group | MDMA-assisted Therapy (100 to 125 mg of MDMA)
Number analyzed (Participants) | 4
score on a scale | -25.00 (2.58)

2. Secondary Outcome: Change From Baseline to Primary Endpoint in Sheehan Disability Scale (SDS for PTSD for MAPS) Total Score
Description: The Sheehan Disability Scale (SDS for PTSD for MAPS) is a self-report assessment of functional impairment. The reporting period for the adapted SDS refers to the past month. The items indicate degree of impairment in the domains of work/school, social life, and home life, with response options based on an eleven-point scale (0=not at all to 10=extremely), with higher scores indicating greater functional impairment.
Time Frame: Baseline (Visit 3) to Primary Endpoint (Visit 19, 18 weeks post-enrollment)
Population: Safety Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MDMA-assisted Therapy (100 to 125 mg of MDMA)
Number analyzed (Participants) | 4
score on a scale
  SDS Total Score at Baseline | 7.4 (1.6)
  SDS Total Score at Primary Endpoint | 2.3 (2.98)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events through study completion (approximately 5 months)
Arm/Group | MDMA-assisted Therapy (100 to 125 mg)
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MDMA-assisted Therapy (100 to 125 mg) (N=4)
Palpitations (Cardiac disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Aphthous ulcer (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Feeling cold (General disorders) | 1
Viral upper respiratory tract infection (General disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 3
Paraesthesia (Nervous system disorders) | 1
Sensory disturbance (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
Aggression (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 3
Depressed mood (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Derealisation (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Nightmare (Psychiatric disorders) | 2
Suicidal ideation (Psychiatric disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Peripheral coldness (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
This was an open-label trial with no placebo comparator in a small sample size (n=4).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-04-02): https://cdn.clinicaltrials.gov/large-docs/87/NCT03485287/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-03): https://cdn.clinicaltrials.gov/large-docs/87/NCT03485287/SAP_003.pdf
  • Informed Consent Form (2018-09-18): https://cdn.clinicaltrials.gov/large-docs/87/NCT03485287/ICF_004.pdf